CLINICAL TRIAL: NCT00867191
Title: A Multi-Centre, Double-Blind, Randomised Comparison Of The Effects Of Desloratadine (Aerius®) And Placebo In The Relief Of Nasal Symptom Scores In Subjects With Seasonal Allergic Rhinitis (Sar) To Cypress Pollen
Brief Title: Comparison of the Effects of Desloratadine and Placebo in the Relief of Nasal Symptom Scores in Subjects With Seasonal Allergic Rhinitis to Cypress Pollen (Study P02836)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P02836
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — desloratadine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Placebo, 1 tablet daily, per os
  Interventions: Drug: Placebo
- 2 (Active Comparator): Desloratadine, one 5 mg tablet daily, per os
  Interventions: Drug: Desloratadine

INTERVENTIONS:
Drug: Placebo — Placebo, 1 tablet daily, per os., 15 days
  Arms: 1
Drug: Desloratadine — Desloratadine, one 5 mg tablet daily, per os, 15 days
  Other Names: SCH 34117
  Arms: 2

SUMMARY:
The purpose of this study was to demonstrate the efficacy (% of change from baseline) of desloratadine to improve the nasal total symptom score of SAR to cypress pollen.

ELIGIBILITY:
Inclusion Criteria:

* Patients must demonstrate their willingness to participate in the study and comply with its procedures by signing a written informed consent.
* Patients must be >=18 years of age, of either gender.
* Women of childbearing potential (includes women who are less than 1 year postmenopausal and women who become sexually active) must be using or agree to use an acceptable method of birth control (e.g. hormonal contraceptive, medically prescribed intrauterine device, condom in combination with spermicide) or be surgically sterilized (e.g. hysterectomy or tubal ligation). Women of childbearing potential who are not currently sexually active must agree and consent to use one of the above-mentioned methods, should they become sexually active while participating in the study.
* Patients must be in good general health; i.e., they must be free of any clinically significant disease (other than SAR to cypress pollen) that could interfere with study evaluations.
* Patients must understand and be able to adhere to the measurement, dosing and visit schedules, and agree to report concomitant medications and adverse events to the investigator or designee.
* Patients must have at least a two-year history (self-reported being acceptable) of intermittent allergic rhinitis specifically from January to March
* Patients must be clinically symptomatic with SAR to cypress pollen at Visit 2 (Day 0): the total (nasal + non-nasal) symptom score must be >=8 with a nasal congestion score >=2. Patients may be rescheduled up to two additional times for the qualifying visit if they do not meet the minimum symptom scores
* A positive skin prick test and / or positive cypress-specific IgE by RAST (>= class 2). These tests should have been performed within 24 months before Visit 1
* Women of childbearing potential must have a negative urine pregnancy test at Visit 2 (Day 0).

Exclusion Criteria:

* Women who are pregnant or nursing.
* Patients who have not observed the designated washout periods for any of the prohibited medications.
* Patients with rhinitis medicamentosa.
* Patients who have had an upper respiratory tract or sinus infection that required antibiotic therapy within 14 days prior to Visit 1 (screening / consent) or patients who have had a viral upper respiratory infection within 7 days prior to Visit 2.
* Patients who have nasal structural abnormalities, including nasal polyps and marked septal deviation, interfering significantly with nasal airflow.
* Patients with a history of hypersensitivity to desloratadine or any of its excipients.
* Patients who are staff personnel directly involved with the administration of this study.
* Patients previously randomised in this study.
* Patients having used any investigational drug in the last 30 days prior to Visit 1.
* Patients who have any current evidence of clinically significant haematopoietic, metabolic, cardiovascular, immunological, neurological, haematological, gastrointestinal, hepatic, renal, psychiatric, cerebrovascular or respiratory disease, or any other disorder which, in the judgment of the investigator, may interfere with the study evaluations or affect patient safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2002-02-01 (Actual); Primary Completion 2003-04-01 (Actual); Study Completion 2003-04-01 (Actual)

PRIMARY OUTCOMES:
The primary objective was to demonstrate the efficacy (as percentage of change from baseline) of desloratadine to improve the nasal total symptom score of SAR to cypress pollen. | After 14 days of treatment

REFERENCES:
- [Derived] Demoly P, Dreyfus I, Dhivert-Donnadieu H, Mesbah K. Desloratadine for the treatment of cypress pollen-induced allergic rhinitis. Ann Allergy Asthma Immunol. 2009 Sep;103(3):260-6. doi: 10.1016/S1081-1206(10)60191-3. PMID 19788025